CLINICAL TRIAL: NCT00243321
Title: Phase I Examination of Combination High Dose-Rate Brachytherapy and/or Intensity Modulated External Beam Therapy for the Comprehensive Local Treatment of Patients With Locally Confined Adenocarcinoma of the Prostate
Brief Title: High Dose-Rate Brachytherapy and/or Intensity Modulated External Beam Radiation Therapy for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-02961
Record Dates: First submitted 2005-10-19; First posted 2005-10-21 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: brachytherapy; intensity-modulated radiation therapy; prostate specific antigen
MeSH Terms: interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HDR brachytherapy -> IMRT (Experimental): Radiotherapy
  Interventions: Procedure: high dose-rate brachytherapy; Procedure: intensity-modulated radiation therapy

INTERVENTIONS:
Procedure: high dose-rate brachytherapy — High dose-rate brachytherapy
Procedure: intensity-modulated radiation therapy — intensity-modulated radiation therapy

SUMMARY:
The principal objective of this study is to demonstrate that patients can safely receive combined High Dose Rate brachytherapy and Intensity-Modulated Radiation Therapy without experiencing a treatment limiting toxicity.

DETAILED DESCRIPTION:
Patients will receive a single High Dose Rate brachytherapy dose of 6 Gy to the prostate, followed by 61 Gy delivered to the prostate and nearby tissues using Intensity-Modulated Radiation Therapy in 28 treatments.

ELIGIBILITY:
Inclusion Criteria:

* TRUS biopsy proven adenocarcinoma of the prostate Pretreatment PSA <30 ng/ml Gleason's sum < 8 clinical stage T1 or T2a,b. patients that are at low-intermediate risk for disease beyond the prostate normal liver function for all patients beginning hormone therapy Karnofsky Performance score > 80 acceptable anesthesia risk as determined through routine pre-operative screening in the VCUHS Diagnostic Testing Clinic

Exclusion Criteria:

* pubic-arch interference or regional disease ( no evidence of metastatic disease for patients whose PSA is greater than 10 ng/ml, Gleason's sum is greater than 6, or T-stage is greater than T2a.

Patients at high risk for distant disease (PSA > 30 ng/ml, Gleason's sum > 8 or clinical stage > T2c), clinically involved seminal vesicles or extension beyond the prostate capsule history of inflammatory bowel disease require steroid or cytotoxic therapy for collagen vascular disease uncontrolled or poorly controlled hypertension uncontrolled or poorly controlled diabetes mellitus history of cancer other than skin cancer within five years of the initiation of protocol treatment history of pelvic irradiation require the routine use of warfarin

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2003-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To demonstrate that patients can safely receive combined HDR brachytherapy and IMRT teletherapy to a total dose consistent with current treatment policies and without experiencing a treatment limiting toxicity | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Hagan, MD, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Background] Amer AM, Mott J, Mackay RI, Williams PC, Livsey J, Logue JP, Hendry JH. Prediction of the benefits from dose-escalated hypofractionated intensity-modulated radiotherapy for prostate cancer. Int J Radiat Oncol Biol Phys. 2003 May 1;56(1):199-207. doi: 10.1016/s0360-3016(03)00086-5. PMID 12694839